CLINICAL TRIAL: NCT05494177
Title: Comparative Study of Premium Monovision and Bilateral Implantation of Trifocal Diffractive Intraocular Lenses
Brief Title: Comparison of Premium Monovision and Bilateral Implantation of Trifocal Diffractive Intraocular Lenses
Status: Completed | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Professor (Associate) of Democritus University of Thrace, Democritus University of Thrace
Other Study IDs: ES13/Th7/07-07-2022
Record Dates: First submitted 2022-08-06; First posted 2022-08-09 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2022-08

CONDITIONS: Presbyopia; Refractive Errors; Cataract
Keywords: pseudophakic presbyopic correction; premium monovision; trifocal diffractive intraocular lenses; extended depth of field intraocular lenses
MeSH Terms: conditions — Presbyopia; Refractive Errors; Cataract | interventions — Contrast Sensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Premium monovision: Patients will undergo to implantation of an extended depth of field intraocular lens in the dominant eye and a trifocal diffractive intraocular lens in the non-dominant eye.
  Interventions: Diagnostic Test: bUDVA, bUIRA, bUNRA, bUICPS, bUNCPS; Diagnostic Test: Contrast sensitivity
- Bilateral trifocal diffractive implantation: Patients will undergo to bilateral implantation of trifocal diffractive lenses.
  Interventions: Diagnostic Test: bUDVA, bUIRA, bUNRA, bUICPS, bUNCPS; Diagnostic Test: Contrast sensitivity

INTERVENTIONS:
Diagnostic Test: bUDVA, bUIRA, bUNRA, bUICPS, bUNCPS — All participants will be assessed on the following clinical indexes:
  1. Binocular uncorrected distant visual acuity (bUDVA) at four meters distance
  2. Binocular uncorrected intermediate reading acuity (bUIRA) at 60 cm
  3. Binocular uncorrected near reading acuity (bUNVA) at 40 cm
  4. Binocular uncorrected intermediate Critical Print Size (bUICPS) at 60 cm
  5. Binocular uncorrected near Critical Print Size (bUNCPS) at 40 cm
  All the above parameters are obtained using the Democritus Digital Acuity & Reading Test (DDART).
Diagnostic Test: Contrast sensitivity — Contrast sensitivity is assessed with the Pelli-Robson test.

SUMMARY:
Primary objective of this study is to compare two presbyopia correction surgical techniques, specificaly premium monovision, in which the dominant eye is corrected with an extended depth of field intraocular lens and the non-dominant eye with a trifocal diffractive intraocular lens, and the bilateral implantation of trifocal diffractive intraocular lenses.

DETAILED DESCRIPTION:
Two study groups will be formed. The first group will include patients who undergone premium monovision and the second will include patients who undergone bilateral implantation of trifocal diffractive intraocular lenses. Patients who have undergone one of the aforementioned categories of presbyopia correction surgery will be selected in order to compare the effectiveness of these techniques by evaluating uncorrected near, intermediate and distant visual acuity, uncorrected Critical Print Size (CPS) in near and intermediate distance, dysphotopic phenomena (glare, halos) through a 4-level severity scale by patients, contrast sensitivity, the need of use glasses for all distances or separately for activities requiring near or distant vision as well as the degree of subjective satisfaction of patient via interview (NEI-VFQ 25). The purpose of measuring these parameters is to calculate, through a mathematical model, the relative effectiveness of each method.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cataract with stage 2 according to the Lens Opacities Classification System III (LOCS-3) grading scale
* Age>45 years

Exclusion Criteria:

* Disability to understand the Greek language and respond to the interview
* Fundus or corneal diseases
* Glaucoma
* Previous intraocular surgery

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were examined at the outpatient of the Department of Ophthalmology of the University General Hospital of Alexandroupolis with the diagnosis of cataract with stage 2 (according to LOCS III) and underwent one of the following presbyopia correction surguries:
  1. Bilateral implantation of trifocal diffractive intraocular lenses
  2. Premium monovision with implantation of an extended depth of focus intraocular lens in the dominant eye and a trifocal diffractive intraocular lens in the non-dominant eye
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Binocular uncorrected distant visual acuity (bUDVA) | 1 year
  bUDVA is obtained using the distance vision test of DDART at four meters distance.
Binocular uncorrected intermediate reading acuity (bUIRA) | 1 year
  bUIRA is obtained using the near vision test of DDART at 60 cm distance.
Binocular uncorrected near reading acuity (bUNRA) | 1 year
  bUNRA is obtained using the near vision test of DDART at 40 cm distance.
Binocular uncorrected intermediate critical print size (bUICPS) | 1 year
  bUICPS is obtained using the near vision test of DDART at 60 cm distance.
Binocular uncorrected near critical print size (bUNCPS) | 1 year
  bUNCPS is obtained using the near vision test of DDART at 40 cm distance.

SECONDARY OUTCOMES:
Dysphotopsia symptoms | 1 year
  Dysphotopsia is evaluated with two direct 4-scale, Likert-type questions (Always, Most of the times, Sometimes, Never) assessing subjective appearance of glare and halos.
Contrast sensitivity | 1 year
  Contrast sensitivity is evaluated with the Pelli-Robson test.
Spectacle independence | 1 year
  Spectacle dependence is assessed for both distant and near vision by two direct 4-scale Likert-type questions (Always, Most of the times, Sometimes, Never).
Subjective satisfaction using Visual Function Index (VF-14) (total score, VF14-Near Vision (NV) score & VF14-Distance Vision (DV) score) | 1 year
  Subjective satisfaction rates are assessed using the prevalent VF-14 questionnaire. Further to the total VF-14 score assessment, two additional scores are calculated: a) Near vision VF score (VF14-NV) derived from items that assess the perceived difficulty in near vision activities (items 1,2,3,7,8,9 and 11), and, b) Distant vision VF score (VF14-DV) derived from items that assess the perceived difficulty of distant vision activities (items 4, 5, 6, 10, 12, 13 and 14).
  VF-14 has a final score from 0 to 100. A score of 100 indicates able to do all applicable activities. A score of 0 indicates unable to do all applicable activities because of vision.

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, MD, PhD, Study Chair — Department of Ophthalmology, University Hospital of Alexandroupolis, Alexandroupolis, Greece
Locations (1):
- Department of Ophthalmology, University Hospital of Alexandroupolis, Alexandroupoli, Evros, Greece

REFERENCES:
- [Derived] Labiris G, Panagis C, Ntonti P, Konstantinidis A, Bakirtzis M. Mix-and-match vs bilateral trifocal and bilateral EDOF intraocular lens implantation: the spline curve battle. J Cataract Refract Surg. 2024 Feb 1;50(2):167-173. doi: 10.1097/j.jcrs.0000000000001336. PMID 37847127